CLINICAL TRIAL: NCT05411874
Title: A Multicenter Randomized Open-label Study of Chidamide Combined With High-dose Dexamethasone Versus High-dose Dexamethasone in the Management of Newly-Diagnosed Immune Thrombocytopenia
Brief Title: A Multicenter Randomized Open-label Study of Chidamide Plus HD-DEX Versus HD-DEX in ITP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Chidamide plus DEX
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Thrombocytopenia
Keywords: HD-DEX; Chidamide
MeSH Terms: conditions — Thrombocytopenia | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chidamide plus HD-DXM (Experimental): Chidamide (orally at 5 mg biw for 24 weeks)
  HD-DXM (orally at 40 mg daily for 4 days)
  Interventions: Drug: Chidamide; Drug: HD-DXM
- HD-DXM (Active Comparator): HD-DXM (orally at 40 mg daily for 4 days )
  Interventions: Drug: HD-DXM

INTERVENTIONS:
Drug: Chidamide — 5mg po biw for 24 weeks
  Arms: Chidamide plus HD-DXM
Drug: HD-DXM — 40mg po qd for 4days

SUMMARY:
Recently, histone deacetylase inhibitors (HDACi) has been used for their anti-inflammatory and immunomodulatory activities. It has been shown that HDACi can alleviate graft-versus-host disease by enhancing the number and function of Foxp3+ Tregs. Our group found that low-dose HDACi alleviated thrombocytopenia in both passive and active murine models of ITP. Furthermore, low-dose HDACi attenuated macrophage phagocytosis of antibody-coated platelets, stimulated production of natural Foxp3+ Tregs, promoted peripheral conversion of T cells into Tregs, and restored Treg suppressive function in vivo and in vitro. The project was undertaking by Qilu Hospital of Shandong University and other 10 well-known hospitals in China. In order to report the efficacy and safety of the low dose chidamide combined with high-dose dexamethasone versus high-dose dexamethasone in the management of ITP.

DETAILED DESCRIPTION:
Primary immune thrombocytopenia (ITP) is an autoimmune bleeding disorder with low platelet count. Low-dose HDACi alleviated thrombocytopenia in both passive and active murine models of ITP. In this multicentre, open-label, randomized controlled trial, newly diagnosed ITP patients will be enrolled from 11 tertiary medical centres in China. Participants will be randomly assigned into the combination group or the monotherapy group by masked statisticians in a 1:1 ratio. The primary endpoints are sustained response at month 6. The secondary outcomes include initial response, time to response, duration of response, bleeding score, health-related quality of life assessment, and safety issue. This study will compare the efficacy and safety of low dose chidamide combined with high-dose dexamethasone versus high-dose dexamethasone monotherapy in adults with primary immune thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed ITP patients need of treatment(s) to minimize the risk of clinically significant bleeding primary ITP confirmed by excluding other supervened causes of thrombocytopenia

Exclusion Criteria:

* pregnancy hypertension cardiovascular disease diabetes liver and kidney function impairment HCV, HIV, HBsAg seropositive status patients with systemic lupus erythematosus and/or antiphospholipid syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Sustained response | 6 month
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up.

SECONDARY OUTCOMES:
Initial response | day 14
  CR: platelet count ≥ 100 × 109/L and absence of bleeding; R: platelet count ≥ 30 × 109/L but < 100 × 109/L and a doubling from baseline and absence of bleeding.
Number of patients with bleeding | 6 month
  Number of patients with bleeding complication. Bleeding symptoms were graded according a standardized bleeding scale specific to primary immune thrombocytopenia on the basis of site and severity of bleeding by Khellaf et al (PMID: 15951296). A modification was made to exclude age from the original scale so that only bleeding symptoms were described. Scores ranged from 0 to 59, with higher values indicating higher bleeding risk.
Number of patients with adverse events | 6 month
  Adverse events were graded according to the Common Terminology Criteria for Adverse Events (version 4.0). At each visit, we recorded adverse events. Routine visits were scheduled once a week for the first 4 weeks and once a month thereafter.
Time to response | 6 month
  The time from starting treatment to time of achievement of CR or R
Duration of response (DOR) | 6 month
  Duration of response was defined as the time from achievement of a complete response or a partial response to the loss of response (platelet count <30 × 10⁹ cells per L; measured on two occasions more than 1 day apart or the presence of bleeding).
Health-related quality of life assessment | 6 month
  Health-related quality of life was assessed using a self-administered immune thrombocytopenia Patient Assessment Questionnaire (ITP-PAQ) at baseline and at week 12. Scores ranged from 0 to 100, with higher values indicating better quality of life.

REFERENCES:
- [Background] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182